CLINICAL TRIAL: NCT06612216
Title: Research on the Scientific Connotation of Cancer Toxin Pathogenesis Based on the Interaction Between Flora and Tumor-Establishment of Cohort Under the Guidance of the Pathogenesis of Cancer Toxin in Traditional Chinese Medicine
Brief Title: Establishment of Cohort Under the Guidance of the Pathogenesis of Cancer Toxin in Traditional Chinese Medicine
Status: Not yet recruiting | Type: Observational
Sponsor: Ying Zhang (Other)
Collaborators: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other); Dongzhimen Hospital, Beijing (Other); Beijing Chest Hospital, Capital Medical University (Other); Shanghai University of Traditional Chinese Medicine (Other); Shaanxi Hospital of Traditional Chinese Medicine (Other); Leling Traditional Chinese Medicine Hospital (Unknown); Henan Medical University (Other)
Responsible Party: Sponsor-Investigator, Ying Zhang, Director, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Other Study IDs: CI2023C025YL
Record Dates: First submitted 2024-09-19; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Cancer
Keywords: flora; microbiota; tumor; cancer toxin
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood, feces, tissue, tongue coating
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- healthy individuals and cancer patients: Comparing the microbiota characteristics of healthy individuals and cancer patients, revealing the differences in microbiota between healthy individuals and cancer patients.
  Interventions: Other: No intervention was carried out
- Patients with different traditional Chinese medicine cancer toxicity syndrome types: According to the classification of traditional Chinese medicine cancer toxin syndrome types, compare the differences in microbiota between the heat toxin syndrome group, dampness toxin syndrome group, stasis toxin syndrome group, phlegm toxin syndrome group, wind toxin syndrome group, and cold toxin syndrome group in cancer patients, and explore the influence of different cancer toxin syndrome types on microbiota composition.
  Interventions: Other: No intervention was carried out
- Patients with different traditional Chinese medicine constitutions: According to the traditional Chinese medicine constitution classification, compare the differences in microbiota among tumor patients with qi stagnation constitution group, phlegm dampness constitution group, damp heat constitution group, blood stasis constitution group, qi deficiency constitution group, yang deficiency constitution group, yin deficiency constitution group, characteristic constitution group, and peaceful constitution group, and explore the influence of different constitution types on the microbiota composition of tumor patients.
  Interventions: Other: No intervention was carried out
- Patients with different tumor burden: Divide tumor patients into tumor bearing group and tumor free group, and explore their microbiota characteristics and differential patterns.
  Interventions: Other: No intervention was carried out
- Patients with different symptom burdens: According to the MDASI Anderson Symptom Scale, compare the differences in microbiota between individuals with mild and severe symptom burdens, and explore the impact of different symptom burdens on the microbiota composition of cancer patients.
  Interventions: Other: No intervention was carried out
- Patients with different treatment and outcome outcomes: Based on the application of different treatment methods and the resulting outcomes in cancer patients, compare the characteristic differences of microbiota between groups and explore the differential expression of microbiota.
  Interventions: Other: No intervention was carried out

INTERVENTIONS:
Other: No intervention was carried out — This study observed differences in microbiota among different groups and therefore did not involve intervention.

SUMMARY:
The study aims to investigate the potential mechanisms by which the interaction between the microbiota and tumors leads to the occurrence and development of cancer by collecting clinical information and biological samples from healthy individuals and cancer patients.

DETAILED DESCRIPTION:
Study Design Types: A prospective, multicenter, observational study.

Observation Content:1.Healthy Individuals:General Information (Demographic Data), Traditional Chinese Medicine Physical Quality Scale, Biological Samples (Fecal, Blood, Tongue Coating, Tongue Appearance Photos, Tissues). 2.Malignant Tumor Patients: General Information (Demographic Data, Disease Information, ECOG Performance Status Score, MDASI Anderson Symptom Inventory), Traditional Chinese Medicine Cancer Toxin Syndrome Scale, Traditional Chinese Medicine Physical Quality Scale, Laboratory and Examination Data, Biological Samples (Fecal, Blood, Tongue Coating, Tongue Appearance Photos, Tissues).

Observation Time Points:1.Healthy Individuals: At the time of enrollment. 2.Malignant Tumor Patients: At the time of enrollment, 1 month after enrollment, every 3 months thereafter until tumor progression.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy individuals:

* Age ≥ 18 years old;
* Informed consent and signed informed consent form.

Inclusion criteria for patients with malignant tumors:

* Patients with malignant tumors diagnosed by pathology or cytology;
* Advanced stage patients who have not received modern medical treatment in the past, or early to mid-stage patients who have completed postoperative radiochemotherapy for ≥ 1 month;
* Age ≥ 18 years old;
* Informed consent and signed informed consent form.

Exclusion Criteria:

Exclusion criteria for healthy individuals:

* Patients with malignant tumors diagnosed by pathology or cytology;
* Those who have taken any antibiotics/probiotics within 1 month before biological sample collection;
* Those with other immune or infectious diseases;
* Those with severe damage to the heart, liver, lungs, or kidney functions;
* Pregnant women, or those with mental illnesses such as depression or schizophrenia;
* Those deemed ineligible for the study by the researcher.

Exclusion criteria for patients with malignant tumors:

* Patients with multiple primary cancers;
* Those who have taken any antibiotics/probiotics within 1 month before biological sample collection;
* Those with other immune or infectious diseases;
* Those with severe damage to the heart, liver, lungs, or kidney functions;
* Pregnant women, or those with mental illnesses such as depression or schizophrenia;
* Those deemed ineligible for the study by the researcher.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy individuals and cancer patients.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-22 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
16S rDNA | 2 years (from enrollment to disease progression).
  16S rDNA detection is a commonly used method in microbial molecular biology for identification and classification of bacteria. It can identify and classify bacteria.

SECONDARY OUTCOMES:
microbiota metagenomics | 2 years (from enrollment to disease progression).
  Metagenomic Sequencing is a technique that studies the total genetic material of all microorganisms in environmental samples. This method does not rely on traditional microbial isolation and cultivation, but instead directly extracts total DNA from environmental samples to obtain new functional genes and bioactive substances by constructing and screening metagenomic libraries.
Untargeted metabolomics | 2 years (from enrollment to disease progression).
  Untargeted Metabolomics is a research method that does not rely on prior knowledge of specific metabolites. Instead, it explores the overall patterns and changes of metabolites by analyzing all detectable metabolites in biological samples.

IPD SHARING:
Plan to Share IPD: No